CLINICAL TRIAL: NCT00933179
Title: A Single-Center, Open-Label, Crossover, Randomized Study to Investigate the Impact of the Transdermal Contraceptive Patch Containing 0.55 mg Ethinylestradiol and 2.1 mg Gestodene (Material no. 80876395) in a 21-day Regimen as Compared to a Monophasic Contraceptive Containing Ethinylestradiol and Levonorgestrel (0.03mg/0.15mg) in a 21-day Regimen on Hemostatic Parameters in 30 Women Aged 18 182 35 Years Over 3 Treatment Cycles in Each Period
Brief Title: FC Patch Low: Metabolism Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 91557; 2008-007024-26 (EudraCT Number)
Record Dates: First submitted 2009-07-03; First posted 2009-07-07 (Estimated); Last update posted 2014-11-14 (Estimated); Status verified 2014-11

CONDITIONS: Contraception
Keywords: Prevention of pregnancy
MeSH Terms: interventions — ethinyl estradiol, levonorgestrel drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: Gestodene/EE Patch (BAY86-5016)
- Arm 2 (Active Comparator)
  Interventions: Drug: EE/Levonorgestrel (Microgynon, BAY86-4977)

INTERVENTIONS:
Drug: Gestodene/EE Patch (BAY86-5016) — 21-day regimen per cycle (1 patch a week for 3 weeks followed by a 7-day patch-free period) for 3 cycles
  Arms: Arm 1
Drug: EE/Levonorgestrel (Microgynon, BAY86-4977) — 21-day regimen per cycle (1 tablet a day for 3 weeks followed by a 7-day tablet-free period) for 3 cycles
  Arms: Arm 2

SUMMARY:
The aim of the present study is to investigate the effects of the transdermal patch on the parameters of hemostasis (blood clotting), lipid (fat), and carbohydrate (sugars) metabolism in healthy women who require contraception.

ELIGIBILITY:
Inclusion Criteria:

* Healthy woman requesting contraception
* Normal cervical smear not requiring further follow-up
* History of regular cyclic menstrual periods
* Willingness to use non-hormonal contraception during the two wash-out cycles both before the start of treatment and between the two treatment periods

Exclusion Criteria:

* Pregnancy or lactation - Obesity (Body Mass Index [BMI] > 30.0 kg/m2)
* Any diseases or conditions that can compromise the function of the body systems
* Any diseases or conditions that might interfere with the conduct of the study or the interpretation of the results
* Any disease or condition that may worsen under hormonal treatment
* Undiagnosed abnormal genital bleeding
* Any medication that could result in excessive accumulation, impaired metabolism, or altered excretion of the study drug or interfere with the conduct of the study or the interpretation of the results

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2009-06; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Prothrombin fragment 1+2, D-dimer | Screening, visit 3-7

SECONDARY OUTCOMES:
Procoagulatory parameters | Screening, visit 3-7
Anticoagulatory parameters | Screening, visit 3-7
Thrombin and Fibrin turnover parameters | Screening, visit 3-7

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Berlin, State of Berlin, Germany

REFERENCES:
- [Result] Junge W, Heger-Mahn D, Trummer D, Merz M. Investigation of the hemostatic effect of a transdermal patch containing 0.55 mg ethinyl estradiol and 2.1 mg gestodene compared with a monophasic oral contraceptive containing 0.03 mg ethinyl estradiol and 0.15 mg levonorgestrel: an open-label, randomized, crossover study. Drugs R D. 2013 Sep;13(3):223-33. doi: 10.1007/s40268-013-0028-2. PMID 24043457
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/